CLINICAL TRIAL: NCT06928467
Title: Primary Care-based Pilot ePCT of an Online Workshop for Family Caregivers of PLWD
Brief Title: Primary Care-based Study of an Online Workshop for Family Caregivers of PLWD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Brown IRB ID: STUDY00000388; U54AG063546 (NIH)
Record Dates: First submitted 2025-04-01; First posted 2025-04-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Family Caregivers; Dementia; Self-management; Depression; Internet-based Intervention
MeSH Terms: conditions — Dementia; Depression

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Principal investigator and biostatistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop (Experimental): A 6-week, online, peer-led small group workshop designed for family caregivers of persons living with dementia.
  Interventions: Behavioral: Building Better Caregivers workshop
- Control (No Intervention): Wait-list control group.

INTERVENTIONS:
Behavioral: Building Better Caregivers workshop — The BBC workshop is a 6-week, online, peer-led small group workshop designed for family caregivers of persons living with dementia or other form of cognitive impairment. It is an evidence-based workshop of the Self-Management Resource Center originally developed at Stanford University for the Veterans Administration and is now licensed for online delivery by Canary Health. Content focuses on increasing participant self-management behaviors, dementia caregiving skills, and peer social support. The workshop uses a peer-facilitated small group format with frequent online interactions between approximately 27 participants on threaded discussion boards. Activities are guided by two trained peer co-facilitators (caregivers themselves). Each week focuses on 2-3 new topics and tools for participants to learn and use. In threaded discussion board conversations participants interact, help each other, and provide peer social support.
  Arms: Workshop

SUMMARY:
Many family and friend caregivers of persons living with dementia experience depression, stress, and other adverse health consequences due to the responsibilities of their caregiving role. These caregivers express a desire for education and support. The overarching goal of this project is to improve education and support for caregivers of persons living with dementia so that they can take better care of themselves and also their person living with dementia.

Building Better Caregivers workshop is an online, 6-week, small group workshop for family caregivers of persons living with dementia that teaches them caregiving skills and how to manage difficult emotions, stress, and other challenging aspects of caregiving. Caregivers also receive support from other caregivers and two trained workshop facilitators and a workbook to keep. The workshop uses asynchronous delivery that allows caregivers to use materials at home when they have time day or night, self-pace their learning, and chat with other caregivers through threaded discussion board conversations.

In this pilot embedded pragmatic clinical trial the investigators will evaluate the workshop among 108 caregivers who receive health care in urban areas of California and rural areas of New York. To achieve the project goals the investigators will (1) determine the feasibility of identifying, enrolling, and randomizing caregivers to a workshop group or wait-list group; (2) assess the feasibility of using electronic health record data as study outcomes, including depressive symptoms of caregivers and emergency room visits and hospitalizations of their patients with dementia; and (3) determine whether caregivers complete the workshop and think it is acceptable.

If this pilot trial is successful, the investigators will have the information necessary to conduct a larger study among many additional caregivers with the long-term goal of improving their health and the well-being of their person with dementia.

DETAILED DESCRIPTION:
The overarching goal of this project is to improve education and support for family caregivers of persons living with dementia so that they can take better care of themselves and also their person living with dementia.

Objectives

The goals of this project are to perform a pilot embedded pragmatic clinical trial (ePCT) of the Building Better Caregivers (BBC) workshop among 108 family caregivers of persons living with dementia (PLWD) receiving care at the University of California San Francisco (UCSF) or Bassett Healthcare Network (Bassett) of New York and, in doing so, pilot test all clinical trial components necessary to the success of a future larger trial. To accomplish these goals, investigators will:

1. Evaluate the feasibility of using pragmatic methods to identify, enroll, and randomize caregivers (N=108) of PLWD who receive healthcare at UCSF or Bassett Healthcare Network to intervention (BBC workshop) or wait-list control group.
2. Determine the feasibility, acceptability, and fidelity of implementing the online 6-week workshop in USCF and Bassett primary care clinics.
3. Assess the feasibility of using pragmatic methods for clinical outcomes ascertainment including caregiver depressive symptoms (primary clinical outcome, collected through usual clinical care approaches) and ER visits and hospitalizations of PLWD (secondary outcomes)

Trial design

The study will use a randomized pilot ePCT design involving 108 family caregivers of PLWD who both receive care within the UCSF or Bassett healthcare systems. Caregivers will be randomized to BBC workshop group or wait-list control group. Outcomes assessors will be blinded to group assignment.

Outcomes

This is a pilot pragmatic randomized controlled trial designed the outcomes focus on feasibility, acceptability and fidelity end points organized by project goals as outlined below:

1. Outcomes to evaluate feasibility of pragmatic methods to identify, enroll, and randomize caregivers

   1. % of invitation letters that are unopened or returned
   2. % of eligible caregivers for whom contact is attempted who enroll
2. Outcomes to determine feasibility, acceptability, and fidelity of implementing workshop

   1. % of caregivers assigned to workshop who complete workshop
   2. % of caregivers assigned to workshop who report the workshop to be acceptable
   3. % of workshop delivered with fidelity (by checklist)
3. Outcomes to assess feasibility of pragmatic methods for clinical outcomes ascertainment

   1. % of enrolled caregivers who complete caregiver depressive symptoms (PHQ-8) survey questions (primary outcome)
   2. emergency room visits and hospitalizations of PLWD (secondary outcomes)

      Study population

      The study population will include 108 family caregivers of PLWD. Caregivers will be patients within the UCSF or Bassett healthcare systems and will be providing support to PLWD receiving primary care at participating UCSF or Bassett clinics. PLWDs partnered with enrolled caregivers will not receive any intervention but their episodes of emergency room (ER) visits or hospitalizations will be extracted from the electronic health record (EHR). The study sites are the UCSF or Bassett healthcare systems and their respective clinics

      Study locations

      The two participating healthcare systems are UCSF and Basset and their respective outpatient clinics.

      Data collection and follow-up

      Baseline data collection occurs in the month prior to cohort launch. Follow-up data collection initiates 3 months after cohort launch and has a 4-week window.

      Intervention

      The BBC workshop is a 6-week, online, peer-led small group workshop designed for family caregivers of persons living with dementia or other form of cognitive impairment. It is an evidence-based workshop of the Self-Management Resource Center originally developed at Stanford University for the Veterans Administration. The intervention is based on Self-Efficacy Theory and has a well-documented protocol that has been applied across multiple preliminary studies. Content focuses on increasing participant self-management behaviors, dementia caregiving skills, and peer social support. The workshop has been demonstrated to improve caregiver depressive symptoms, stress, self-efficacy, and well-being and reduce emergency department visits and hospitalizations of their PLWDs. The workshop uses a peer-facilitated small group format with frequent online interactions between approximately 27 participants on threaded discussion boards. Activities are guided by two trained peer co-facilitators (caregivers themselves). Participants use screen names to protect their anonymity, if desired. Each week, participants are asked to log on at least 2-3 times a week for about 10 to 30 minutes at a time. The workshop can be accessed with lower speed internet (e.g., no need for broadband) and at any time of day or night. Participation does not require "real time" attendance or video (e.g., Zoom). Instead, caregivers interact in group conversations by posting on discussion boards. Each week focuses on 2-3 new topics and tools for participants to learn and use. Participants answer questions about their caregiving challenges and their responses are posted for everyone to see. In threaded discussion board conversations participants interact, help each other, and provide peer social support. Canary Health is the digital health company that holds the license from the Self-Management Resource Center to deliver the online version of the workshop on its online platform.

      Randomization and blinding

      The study requires approximately 36 caregivers per study cohort and 3 cohorts (108 total caregiver participants). The study will use a randomization ratio of 3:1 to assign approximately 27 to workshop and 9 to wait-list control. This randomization approach enables faster accrual for each cohort. Interested wait-list control group caregivers also will be offered the workshop after their 3-month trial participation is completed.

      Inclusion and exclusion criteria

      These criteria are described elsewhere on clinicaltrials.gov.

      Data analysis and statistical considerations

      This pilot study is not powered to determine effectiveness of the workshop. Instead, we use statistical assessment and a CI-based approach to establish progression criteria for proceeding to a future large ePCT the following endpoints: feasibility of workshop completion by caregivers, workshop acceptability to caregivers, and feasibility of clinical outcome ascertainment of PHQ-8 depression symptoms score (primary clinical outcome). The Table indicates the possible scenarios we will use to decide whether a full ePCT is warranted. For each feasibility endpoint we identify possible observed outcomes and a CI approach that identifies a lower bound for the criteria (green, yellow, red) for proceeding to a future larger ePCT. Meeting the "green" criteria indicates to move forward to a future larger ePCT (based on that criterion); "yellow" indicates possibly move forward (but consider necessary modifications, e.g., intervention tailoring to particular sub-groups/settings); and " red" indicates do not move forward.
      1. Feasibility of workshop completion

         Green: Completion rate 75%, 95% CI between (65%, 85%) with a probability of 0.942, Lower bound is 65%

         Yellow: Completion rate 65%, 95% CI between (54.4%, 75.6%) with a probability of 0.970, Lower bound is 54%

         Red: Completion rate <54%
      2. Acceptability of workshop

         Green: Completion rate 75%, 95% CI between (65%, 85%) with a probability of 0.942, Lower bound is 65%

         Yellow: Completion rate 65%, 95% CI between (54.4%, 75.6%) with a probability of 0.970, Lower bound is 54%

         Red: Completion rate <54%
      3. Feasibility of outcome ascertainment (PHQ-8)

      Green: Outcome ascertainment 74%, 95% CI between (65%, 83%) with a probability of 0.996, Lower bound is 65%

      Yellow: Outcome ascertainment 65%, 95% CI between (55.8%, 74.2%) with a probability of 0.973, Lower bound is 56%

      Red: Outcome ascertainment <56%

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older (no upper limit)
* Sex/Gender: any sex, any gender
* Race/ethnicity: any race/ethnicity
* Able to read and write in English
* Have internet access on any device (computer, tablet, smartphone) but does not require high speed internet
* Provide care to a person living with dementia who is a primary care patient participating health system, i.e., UCSF or Bassett
* Receive own healthcare at participating health system, i.e., UCSF or Bassett

Exclusion Criteria:

- Investigator discretion for clinical safety or protocol adherence reasons, e.g., potential participant who might not be able to meet the time requirements of the study (anticipating a move)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
3a. Percent of enrolled caregivers who complete caregiver depressive symptoms (PHQ-8) survey questions | Up to 4 months
  Percentage of enrolled caregivers who complete caregiver depressive symptoms survey questions from the 8-item Patient Health Questionnaire (PHQ-8), with score range 0-24 (higher score indicates worse depressive symptoms), with range 0% to 100% (higher percentage indicates higher completion rate).

SECONDARY OUTCOMES:
3b. Healthcare utilization of emergency room visits and hospitalizations by person living with dementia | Up to 5.5 months
  Healthcare utilization days measured as emergency room and hospitalization days of use among persons living with dementia who are care partners of enrolled caregivers during the 3-month post-group delivery period, with range 0-90 days (higher count indicates more days).

OTHER OUTCOMES:
1a. Percent of invitation letters that are unread | Baseline
  Percentage of invitation letters that are unread, with unread defined as being unopened electronic messages in the electronic health record or returned paper letters returned by US postal service), with range 0% to 100% (higher percentage indicates higher unread rate).
1b. Percent of eligible caregivers for whom contact is attempted who enroll | Baseline
  Among caregivers for whom contact is attempted by invitation letter, the percentage of caregivers who enroll, with range 0% to 100% (higher percentage indicates higher enrollment rate).
2a. Percent of caregivers assigned to workshop who complete workshop | Up to 6 weeks
  Among caregivers who are assigned to workshop, the percentage of caregivers who complete the workshop, with range 0% to 100% (higher percentage indicates higher completion rate).
2b. Percent of caregivers assigned to workshop who report the workshop to be acceptable based on likelihood to recommend to others | Up to 4 months
  Among caregivers who are assigned to workshop, the percentage of caregivers who report the workshop to be acceptable using a likelihood to recommend 10-point Likert scale, with range 0 to 10 and scale anchors at each end, with 0 anchored by "not at all likely" and 10 anchored by "extremely likely" (higher score indicates higher acceptability).
2c. Percent of workshop delivered with fidelity (by checklist) | Up to 6 weeks
  Among workshops, percentage of delivery weeks that meet all elements of fidelity checklist for that week, with range 0% to 100% (higher percentage indicates greater delivery fidelity).

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Yank, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - The Mary Imogene Bassett Hospital dba Bassett Medical Center-Bassett Healthcare Network, Cooperstown, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorig K, Thompson-Gallagher D, Traylor L, et al. Building Better Caregivers: a pilot online support workshop for family caregivers of cognitively impaired adults. Journal of applied gerontology. 2012;31 423-437.
- [Background] Santoyo-Olsson J, Lorig K, Romo EM, Luzanilla M, Ramirez GA, Cheng J, Chesla C, Covinsky KE, Karliner L, Thompson DG, Fahrenwald N, Yank V. Study protocol for a hybrid effectiveness-implementation trial of the Building Better Caregivers online workshop for rural family/friend caregivers of people living with dementia. Contemp Clin Trials. 2022 Oct;121:106903. doi: 10.1016/j.cct.2022.106903. Epub 2022 Aug 31. PMID 36057375
- [Background] Yank V, Gale RC, Nevedal A, Okwara L, Koenig CJ, Trivedi RB, Dupke NJ, Kabat M, Asch SM. Improving Uptake of a National Web-Based Psychoeducational Workshop for Informal Caregivers of Veterans: Mixed Methods Implementation Evaluation. J Med Internet Res. 2021 Jan 7;23(1):e16495. doi: 10.2196/16495. PMID 33410759
- [Background] Lorig K, Ritter PL, Laurent DD, Yank V. Building Better Caregivers: A Pragmatic 12-Month Trial of a Community-Based Workshop for Caregivers of Cognitively Impaired Adults. J Appl Gerontol. 2019 Sep;38(9):1228-1252. doi: 10.1177/0733464817741682. Epub 2017 Nov 14. PMID 29165000
- [Background] 2023 Alzheimer's disease facts and figures. Alzheimers Dement. 2023 Apr;19(4):1598-1695. doi: 10.1002/alz.13016. Epub 2023 Mar 14. PMID 36918389